CLINICAL TRIAL: NCT01296854
Title: The Effect of Spa Treatment on Chronic Obstructive Pulmonary Disease
Acronym: BPCeaux
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The feasability of inclusions has proven very low.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2010/NM-02; 2010-A00693-36 (Other: RCB number)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: spa therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (No Intervention): The patients randomized into this arm of the study will not have spa therapy.
- Spa Therapy (Experimental): The patients randomized into this arm of the study will have 3 weeks of spa therapy
  Interventions: Other: Spa therapy

INTERVENTIONS:
Other: Spa therapy — 3 weeks of spa therapy
  Arms: Spa Therapy

SUMMARY:
The primary objective of this study is to measure and compare the number of exacerbations (moderate or severe) between the two groups of randomized patients with and without thermal treatment). An exacerbation is defined by an increase in symptoms which justifies a unscheduled medical action: increased daily treatment and / or use of corticosteroids, and / or antibiotic therapy. Exacerbations are documented via prescriptions, hospitalisation reports or unscheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient must have chronic obstructive pulmonary disease
* Obstructive ventilation problem: Tiffeneau index (expiratory volume in one second / slow vital capacity) < 70%
* Expiratory volume in one second < 80% of the theoretical value
* Reversibility < 12% after inhalation of bronchodilators
* Smokers or ex smokers
* Available for study monitoring
* Has access to diagnostic, medical and therapeutic care according to the best, current criteria (see the recommendations of the French Language Pseumologist Society)

Exclusion Criteria:

* The patient is participating in another study
* The patient has participated in another study in the past 12 months
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is in military service (unavailable for monitoring)
* Patient is on parole or otherwise has their liberty restricted by administrative or judiciary decision
* The patient is pregnant, or does not have contraception
* The patient is breastfeeding
* Patient has neoplastic disease
* Patient has asthma
* Patient has another, evolving pulmonary disease (tuberculosis, pulmonary interstitium disease, active or recent pulmonary infection)
* Patient has a clinical history indicating asthma or another respiratory disease (in particular bronchiectasis, pneumoconiosis and other occupational diseases, history of pulmonary neoplasia, HIV, immunosuppressive therapy including corticosteroids in the long term
* Patient has respiratory insufficiency
* Hypereosinophilic patient (the number of polynuclear eosinophils is > 0.5 giga/l; confirmed on 2 hemograms)
* Recent psychiatric trouble (less than 1 year)
* Takes illegal drugs
* Patient does not have pneumological care according to the standards set by the French Language Pneumologist Society

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations | 12 months after the beginning of treatment
  Exacerbation = increase in symptoms (IS) justifying an unprogrammed therapeutic intervention (TI). An IS = increase in >=2 of the following minor symptoms for >= 2 consecutive days (CD): (i) dyspnea, (ii) volume or (iii) purulence of sputum. Or an increase in any 1 of the following major symptoms associated with any of the minor symptoms for at least 2 CD: (a) sore throat, (b) cold, (c) fever, (d) coughing, (e) wheezing. A TI = systemic corticoids and/or antibiotics. An exacerbation is defined as severe if TI is accompanied by a hospital stay > 24h, and as "moderate" otherwise.

SECONDARY OUTCOMES:
change in the BODE score | 3 weeks
change in SF36 questionnaire scores | 3 weeks
  the SF36 quality of life questionnaire
Cost (€) | 3 weeks
  Costs are evaluated from the point of view of payers associated with the pathology.
C reactive protein (mg/l) | 3 weeks
  blood work
Eosiniphil count (thou/ml) | 3 weeks
  blood work
Number of exacerbations | 3 weeks
  Exacerbation = increase in symptoms (IS) justifying an unprogrammed therapeutic intervention (TI). An IS = increase in >=2 of the following minor symptoms for >= 2 consecutive days (CD): (i) dyspnea, (ii) volume or (iii) purulence of sputum. Or an increase in any 1 of the following major symptoms associated with any of the minor symptoms for at least 2 CD: (a) sore throat, (b) cold, (c) fever, (d) coughing, (e) wheezing. A TI = systemic corticoids and/or antibiotics. An exacerbation is defined as severe if TI is accompanied by a hospital stay > 24h, and as "moderate" otherwise.
change in the BODE score | 3 months
change in the BODE score | 6 months
change in the BODE score | 9 months
change in the BODE score | 12 months
change in SF36 questionnaire scores | 3 months
  the SF36 quality of life questionnaire
change in SF36 questionnaire scores | 6 months
  the SF36 quality of life questionnaire
change in SF36 questionnaire scores | 9 months
  the SF36 quality of life questionnaire
change in SF36 questionnaire scores | 12 months
  the SF36 quality of life questionnaire
Cost (€) | 3 months
  Costs are evaluated from the point of view of payers associated with the pathology.
Cost (€) | 6 months
  Costs are evaluated from the point of view of payers associated with the pathology.
Cost (€) | 9 months
  Costs are evaluated from the point of view of payers associated with the pathology.
Cost (€) | 12 months
  Costs are evaluated from the point of view of payers associated with the pathology.
Number of exacerbations | 3 months
  Exacerbation = increase in symptoms (IS) justifying an unprogrammed therapeutic intervention (TI). An IS = increase in >=2 of the following minor symptoms for >= 2 consecutive days (CD): (i) dyspnea, (ii) volume or (iii) purulence of sputum. Or an increase in any 1 of the following major symptoms associated with any of the minor symptoms for at least 2 CD: (a) sore throat, (b) cold, (c) fever, (d) coughing, (e) wheezing. A TI = systemic corticoids and/or antibiotics. An exacerbation is defined as severe if TI is accompanied by a hospital stay > 24h, and as "moderate" otherwise.
Number of exacerbations | 6 months
  Exacerbation = increase in symptoms (IS) justifying an unprogrammed therapeutic intervention (TI). An IS = increase in >=2 of the following minor symptoms for >= 2 consecutive days (CD): (i) dyspnea, (ii) volume or (iii) purulence of sputum. Or an increase in any 1 of the following major symptoms associated with any of the minor symptoms for at least 2 CD: (a) sore throat, (b) cold, (c) fever, (d) coughing, (e) wheezing. A TI = systemic corticoids and/or antibiotics. An exacerbation is defined as severe if TI is accompanied by a hospital stay > 24h, and as "moderate" otherwise.
Number of exacerbations | 9 months
  Exacerbation = increase in symptoms (IS) justifying an unprogrammed therapeutic intervention (TI). An IS = increase in >=2 of the following minor symptoms for >= 2 consecutive days (CD): (i) dyspnea, (ii) volume or (iii) purulence of sputum. Or an increase in any 1 of the following major symptoms associated with any of the minor symptoms for at least 2 CD: (a) sore throat, (b) cold, (c) fever, (d) coughing, (e) wheezing. A TI = systemic corticoids and/or antibiotics. An exacerbation is defined as severe if TI is accompanied by a hospital stay > 24h, and as "moderate" otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Molinari, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes; Jean Victor Hérété, MD, Principal Investigator — Amélie les Bains
Locations (6):
- France (6):
  - Private practice: Karim Berkani, Aix-les-Bains
  - Private practice: Jean Hérété, Amélie Les Bains Palalda
  - Private practice: Pierre Ethève, Briey
  - Private practice: Marc Bellier, Ceret
  - Private practice: Pierre Olivier, Perpignan
  - Private practice: Muriel Nouvelle, Saint-Amand-les-Eaux